CLINICAL TRIAL: NCT00167583
Title: Phase III Study of Recombinant Human Interferon-alpha2a Versus Cyclosporin A for the Treatment of Ocular Behcet's Disease - a National,Randomised, Single-masked Controlled Trial (INCYTOB)
Brief Title: Interferon-alpha2a Versus Cyclosporin A for Severe Ocular Behcet's Disease (INCYTOB)
Acronym: INCYTOB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKF 105-0-0; BMBF-01KG0706 (Other Grant/Funding Number: German Ministry of Health)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2016-05

CONDITIONS: Behcet's Disease; Panuveitis; Posterior Uveitis; Retinal Vasculitis
Keywords: Ocular Behcet's disease; Panuveitis; Posterior Uveitis; Retinal vasculitis; Treatment; Interferon-alpha; Cyclosporin A
MeSH Terms: conditions — Behcet Syndrome; Panuveitis; Uveitis, Posterior; Retinal Vasculitis | interventions — Cyclosporine; Interferon alpha-2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Cyclosporin A (Active Comparator): Cyclosporin A
  Interventions: Drug: Cyclosporin A
- B Interferon alpha (Active Comparator): Interferon-alpha2a
  Interventions: Drug: Interferon-alpha2a

INTERVENTIONS:
Drug: Cyclosporin A — 3 mg/kg bw, augmented to 5 mg if necessary and combined with prednisolone. Adapted to serum levels
  Other Names: Sandimmun neoral
  Arms: A Cyclosporin A
Drug: Interferon-alpha2a — 3-6 million iU per day sc., augmented to up to 9 if necessary, later reduced (according to clinical response) to 3 x 3 million iU /week.
  Other Names: Roferon
  Arms: B Interferon alpha

SUMMARY:
The purpose of this study is to investigate if interferon-alpha2a is superior to the standard treatment with cyclosporin A for the treatment of severe ocular manifestations of Behcet's disease.

DETAILED DESCRIPTION:
Behcet's disease is a multisystem vasculitis often involving ocular (retinal) blood vessels (in 70% of all cases). This form of uveitis or retinal vasculitis still leads to blindness in 25 to 50% of the patients irrespective of immunosuppressive treatment.

The aim of the study is to evaluate if Interferon-alpha2a is superior to the present standard treatment (cyclosporin A (CSA)) for severe ocular (panuveitis, posterior uveitis, retinal vasculitis) Behçet's Disease (BD) and significantly improves visual prognosis and quality of health and life of the patients with ocular BD and is acting more rapidly than standard treatment. Furthermore, we want to evaluate if IFN-α induces long term remissions of ocular BD which can be maintained without further medical treatment.

The patients are randomised into two treatment groups (IFN/CSA) and treated for one year according to an algorithm which adapts dosages to clinical course. A crossover from one treatment arm to the other is planned in case of inefficacy.

ELIGIBILITY:
Inclusion Criteria:

* Behçet's disease fulfilling the International Study Group Criteria with active pan- or posterior uveitis (according to the posterior uveitis scoring system) or retinal vasculitis and active disease according to the Behcet's Disease activity scoring system.

Exclusion Criteria:

* Previous treatment with interferon-α or cyclosporin A
* Pregnancy, breast feeding women, malignancy
* Renal impairment (creatinine > 1.5 mg/dl)
* Uncontrolled hypertension or diabetes
* Depression or other psychic disorders(also history of depression)
* History of acute or chronic inflammatory joint or autoimmune disease
* Organ or bone marrow transplant recipient, cardiac failure > NYHAIII
* Acute liver disease with SGPT 2x above normal
* White blood cell count < 3500/mm3
* Platelet count < 100000/mm3
* Hgb < 8.5g/dl
* Body weight <45 kg
* Alcohol abuse or drug abuse
* Mental impairment
* Uncooperative attitude

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvement of disease activity and preservation of visual acuity (monthly, at one and 2 years) | 2 years
Time to improvement and remission | 2 years

SECONDARY OUTCOMES:
Laboratory values for inflammatory activity (monthly) | 2 years
Number of switches from one treatment to the other | 2 years
Quality of life for patients with low vision (monthly) | 2 years
Number of ocular and non-ocular relapses (1 year, 2 years) | 2 years
Duration of the treatment-free period (second year) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ina Koetter, MD, Principal Investigator — Tuebingen University Hospital
Locations (1):
- Department of Internal Medicine II and Department of Ophthalmology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kotter I, Gunaydin I, Zierhut M, Stubiger N. The use of interferon alpha in Behcet disease: review of the literature. Semin Arthritis Rheum. 2004 Apr;33(5):320-35. doi: 10.1016/j.semarthrit.2003.09.010. PMID 15079763
- [Background] Kotter I, Vonthein R, Zierhut M, Eckstein AK, Ness T, Gunaydin I, Grimbacher B, Blaschke S, Peter HH, Stubiger N. Differential efficacy of human recombinant interferon-alpha2a on ocular and extraocular manifestations of Behcet disease: results of an open 4-center trial. Semin Arthritis Rheum. 2004 Apr;33(5):311-9. doi: 10.1016/j.semarthrit.2003.09.005. PMID 15079762
- [Background] Kotter I, Zierhut M, Eckstein AK, Vonthein R, Ness T, Gunaydin I, Grimbacher B, Blaschke S, Meyer-Riemann W, Peter HH, Stubiger N. Human recombinant interferon alfa-2a for the treatment of Behcet's disease with sight threatening posterior or panuveitis. Br J Ophthalmol. 2003 Apr;87(4):423-31. doi: 10.1136/bjo.87.4.423. PMID 12642304
- [Background] Stuebiger N, Koetter I, Zierhut M. Complete regression of retinal neovascularization after therapy with interferon alfa in Behcet's disease. Br J Ophthalmol. 2000 Dec;84(12):1437-8. doi: 10.1136/bjo.84.12.1432g. No abstract available. PMID 11186866
- [Background] Kotter I, Aepinus C, Graepler F, Gartner V, Eckstein AK, Stubiger N, Kaskas B, Zierhut M, Bultmann B, Kandolf R, Kanz L. HHV8 associated Kaposi's sarcoma during triple immunosuppressive treatment with cyclosporin A, azathioprine, and prednisolone for ocular Behcet's disease and complete remission of both disorders with interferon alpha. Ann Rheum Dis. 2001 Jan;60(1):83-6. doi: 10.1136/ard.60.1.83. No abstract available. PMID 11114291
- [Background] Deuter CM, Kotter I, Gunaydin I, Zierhut M, Stubiger N. [Ocular involvement in Behcet's disease: first 5-year-results for visual development after treatment with interferon alfa-2a]. Ophthalmologe. 2004 Feb;101(2):129-34. doi: 10.1007/s00347-003-0927-7. German. PMID 14991308
- [Background] Kotter I, Deuter C, Stubiger N, Zierhut M. Interferon-a (IFN-a) application versus tumor necrosis factor-a antagonism for ocular Behcet's disease: focusing more on IFN. J Rheumatol. 2005 Aug;32(8):1633; author reply 1634. No abstract available. PMID 16078350
- See also: Homepage with informations on Behcet's Disease and on the study protocol , treatment algorithms and centres (in German) — http://www.medizin.uni-tuebingen.de/webim2/ifa1.htm